CLINICAL TRIAL: NCT00357695
Title: Role of the Parieto-Frontal Network in Automatic Processing of Visually Presented Objects
Brief Title: Role of the Brain in Processing Visually Presented Objects
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040047; 04-N-0047
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-28

CONDITIONS: Healthy; Motor Skills
Keywords: Praxis; Grasping; Premotor Cortex; Visuo-Motor Integration; Motor Imagination

SUMMARY:
This study will examine the parts of the brain that use visual information to perform movements. Patients with certain brain lesions tend to have difficulty in processing visually presented objects. This study will look at the brain mechanisms underlying the visuo-motor integration.

Healthy normal volunteers between 20 and 60 years of age are eligible for this study. People who have had a severe head injury with loss of consciousness or any other mental or neurological disorder diagnosed by a doctor may not participate. Candidates will be screened with a medical history, a physical examination focusing on finger movements, and a questionnaire.

Participants' brain activity will be recorded using two techniques - magnetoencephalography(MEG) and magnetic resonance imaging (MRI) - while they watch pictures of various objects flashed on a screen. MEG is a procedure to record magnetic field changes produced by brain activity. During the recording, the subject sits comfortably in an armchair in a dimly lit room and watches pictures presented on a screen. About 50 pictures are shown per session. There are about five sessions, separated by 3-minute breaks. Functional MRI involves taking pictures of the brain using MRI while the subject performs a task. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The MRI scanner is a metal cylinder surrounded by a magnetic field. The subject lies still on a table that can slide in and out of the scanner. During the scan, he or she looks at pictures in six test blocks of 1 minute each, with 30-second breaks between blocks.

DETAILED DESCRIPTION:
Objectives: Patients with frontal lobe lesions tend to grasp visually presented objects automatically and forcefully (forced grasping). Grasping of a milder form is seen in infants and the aged population. These facts suggest the presence of an inherent mechanism for suppressing the automatic tendency toward grasping in the healthy adult brain. Previous studies suggest that the parieto-frontal network, especially the lateral premotor cortex, play a role in the cognition of graspable objects and execution of reaching/grasping. Although the task of reaching/grasping in human beings has been studied mainly by neuroimaging techniques, its cognitive and executive aspects have not been clearly distinguished. Therefore, this project aims to elucidate the mechanisms underlying 'automatic grasping' in humans, focusing on the perceptive/cognitive aspect of the reaching/grasping movements.

Study population and design: Pictures of graspable objects and non-graspable objects are visually presented to 45 healthy adult volunteers. Since this study aims to clarify the mechanism of the human brain for automatically recognizing graspable objects, part of this study will require no response task. Additionally, in order to assess how the automatic functions compare to overt mechanisms, an extra testing session will explore making overt judgments of the pictures.

Outcome measures: The brain activations are investigated by event-related magnetic fields, which have high temporal resolution, and by event-related functional magnetic resonance imaging (fMRI), which has relatively high spatial resolution. It is expected that the lateral premotor cortex, in addition to the parietal cortex, is activated by the visual presentation of graspable objects at a shorter latency, and more strongly, as compared with non-graspable objects, even without any actual motor tasks to follow. Additionally, overt grasping of graspable objects will involve similar areas.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy male or female subjects between the ages of 20 and 60 years old will be eligible within the limits of the exclusion criteria below.

EXCLUSION CRITERIA:

A previous history of neurological diseases will be carefully taken by direct interview by the Principal or Associate Investigators. Subjects who had a head injury (severe enough to cause loss of consciousness) or other brain diseases causing mental disturbance, sensory impairment, or motor dysfunction in the past will be excluded. Subjects who have metals either in the mouth, such as dental prostheses, or in the head, such as surgical clips from any previous surgical procedures, are also excluded due to technical limitations in terms of MEG. Furthermore, subjects wearing glasses for visual correction and those with poor vision, even with contact lenses, are excluded also due to technical limitations for MEG. Subjects who have pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments, and welders and metal workers are excluded for MRI for the sake of safety of subjects. Finally, by doing a brief neurological examination of finger movements, the subjects with poor performance of fine finger movements or those who are judged to have mirror movements will be excluded.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Start 2003-11-18; Study Completion 2008-10-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jeannerod M, Arbib MA, Rizzolatti G, Sakata H. Grasping objects: the cortical mechanisms of visuomotor transformation. Trends Neurosci. 1995 Jul;18(7):314-20. PMID 7571012
- [Background] Chan JL, Ross ED. Alien hand syndrome: influence of neglect on the clinical presentation of frontal and callosal variants. Cortex. 1997 Jun;33(2):287-99. doi: 10.1016/s0010-9452(08)70005-4. PMID 9220259
- [Background] Jeannerod M, Decety J, Michel F. Impairment of grasping movements following a bilateral posterior parietal lesion. Neuropsychologia. 1994 Apr;32(4):369-80. doi: 10.1016/0028-3932(94)90084-1. PMID 8047246